CLINICAL TRIAL: NCT02773433
Title: Proportional Assist Ventilation Versus Volume-Assist-Control After a Failed Spontaneous Breathing Trial: a Randomized Controlled Trial
Brief Title: PAV vs Assist Control After Failed SBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rodrigo Cavallazzi, Assistant Professor of Medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.1009
Record Dates: First submitted 2016-05-12; First posted 2016-05-16 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Weaning Mode Comparison
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAV group (Experimental): Using Proportional Assist Ventilation after failed Spontaneous Breathing Trial
  Interventions: Other: Proportional Assist Ventilation
- Control group (No Intervention): Using Volume Assist Control mode after failed SBT

INTERVENTIONS:
Other: Proportional Assist Ventilation
  Other Names: PAV
  Arms: PAV group

SUMMARY:
The primary aim of this research is to determine the feasibility of conducting a randomized controlled trial comparing two ventilation modes in patients admitted to the ICU who require mechanical ventilation. The investigators plan to include patients on mechanical ventilation with low support (PaO2/FiO2 ratio > 200, FiO2 < 0.5 and PEEP < 8) for a period no longer than 48 hrs. There are a number of potential barriers to enroll patients in the study. Importantly patients will have to be enrolled within 48 hours from the time they meet inclusion criteria.

The secondary aims are to determine the impact of proportional assist-ventilation (PAV) versus volume assist-control (VAC) ventilation by evaluating the number of ventilation-free days, development of Intensive Care Unit (ICU) delirium, use of sedative/ analgesic medications, use of antipsychotic medications, length of stay in the intensive care unit and hospital, reintubations within 24 hours, adverse events, and mortality in the two groups of patients.

DETAILED DESCRIPTION:
Overview of Design Randomized controlled pilot study comparing mechanical ventilation modes and daily spontaneous trial combination, in patients requiring invasive mechanical ventilation with low ventilator support (PaO2/Fio2 ratio > 200, FiO2 < 0.5 & PEEP <8) for a period not greater than 48 hrs.

Hypothesis The investigators hypothesize that 50 % of patients approached will agree to enrollment in this clinical trial over a period of 4 months. The investigators hypothesize 80% of the patients meeting inclusion criteria will be approached in a timely manner. The investigators also propose that PAV mode ventilation will be superior to ACV based on clinical outcome measurements.

Study Subjects Consecutive adult patients requiring invasive mechanical ventilation on low ventilator support (as mentioned above) for a period not greater than 48 hrs will be enrolled if they or their proxy consent for the study. The study will be performed in the intensive care units of University of Louisville and Jewish Hospital in Louisville, KY.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 yrs old
2. Patient or proxy available in the hospital to consent
3. Receipt of invasive mechanical ventilation on low ventilator support (Po2/Fio2 ratio >200, Fio2 <60% & PEEP <8) for a period not greater than 48 hrs

Exclusion Criteria:

1. Pregnant patients
2. Terminal diseases (e.g. advanced or metastatic malignancy, liver cirrhosis with an estimated 3 month mortality > 50%)
3. Severely depressed respiratory drive
4. Receipt of neuromuscular blocker
5. Bronchopleural fistula
6. Inability to obtain consent from patients or their proxies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
proportion of patients who meet criteria for enrollment who are approached in a timely manner | 1 year
patient enrollment number over time | 1 year
compliance with the ventilator settings | 1 year

SECONDARY OUTCOMES:
Ventilation free days from the time patient is enrolled in the study | 1 year
Development of ICU delirium Based on CAM ICU | 1 year
Use of sedative or analgesic medications | 1 year
Use of antipsychotic medications | 1 year
Reintubations within 24 hrs | 1 year
Length of stay in the intensive care unit | 1 year
Length of stay in the hospital | 1 year
Adverse events | 1 year
In hospital mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Cavallazzi, MD, Principal Investigator — University of Louisville
Locations (1):
- UofLouisville, Louisville, Kentucky, United States